CLINICAL TRIAL: NCT04482309
Title: A Phase 2, Multicenter, Open-label Study to Evaluate the Efficacy and Safety of Trastuzumab Deruxtecan (T-DXd, DS-8201a) for the Treatment of Selected HER2 Expressing Tumors (DESTINY-PanTumor02)
Brief Title: A Phase 2 Study of T-DXd in Patients With Selected HER2 Expressing Tumors
Acronym: DPT02
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D967VC00001; 2023-504721-39-02 (Registry Identifier: EU CTIS); 2020-001574-29 (EudraCT Number)
Record Dates: First submitted 2020-07-20; First posted 2020-07-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Part 1: Bladder, Biliary Tract, Cervical, Endometrial, Ovarian, Pancreatic Cancer, Rare Tumors, Any Tumor Type Excluding Breast, Gastric, Colorectal Cancer; Part 2: HER2 Expressing/Amplified Solid Tumors Excluding Breast, Gastric, Colorectal Cancer
Keywords: T-DXd, DS-8201a, Trastuzumab Deruxtecan, HER2
MeSH Terms: conditions — Pancreatic Neoplasms; Colorectal Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Intervention Model Description: This study will consist of Part 1 which includes 7 cohorts of: urothelial bladder cancer, biliary tract cancer, cervical cancer, endometrial cancer, ovarian cancer, pancreatic cancer, and rare tumors; and Part 2 which includes 5 cohorts A to E of: A) any tumor type that is HER2 IHC 3+ (excluding breast, gastric cancer, and colorectal cancer), B) any tumor type that is HER2 IHC 2+/ISH+ (excluding breast, gastric cancer, and colorectal cancer), C) HER2 IHC 2+ or 1+ endometrial cancer, D) HER2 IHC 2+ or 1+ ovarian cancer, and E) HER2 IHC 2+ or 1+ cervical cancer.
Masking Description: This study is Open-Label Study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Part 1 Cohort 1 (Experimental): Biliary tract cancer
  Interventions: Drug: Trastuzumab deruxtecan
- Part 1 Cohort 2 (Experimental): Bladder cancer
  Interventions: Drug: Trastuzumab deruxtecan
- Part 1 Cohort 3 (Experimental): Cervical cancer
  Interventions: Drug: Trastuzumab deruxtecan
- Part 1 Cohort 4 (Experimental): Endometrial cancer
  Interventions: Drug: Trastuzumab deruxtecan
- Part 1 Cohort 5 (Experimental): Ovarian cancer
  Interventions: Drug: Trastuzumab deruxtecan
- Part 1 Cohort 6 (Experimental): Pancreatic cancer
  Interventions: Drug: Trastuzumab deruxtecan
- Part 1 Cohort 7 (Experimental): Rare tumors
  Interventions: Drug: Trastuzumab deruxtecan
- Part 2 Cohort A (Experimental): Any tumor type that is HER2 IHC 3+ (excluding breast, gastric cancer, and colorectal cancer)
  Interventions: Drug: Trastuzumab deruxtecan
- Part 2 Cohort B (Experimental): Any tumor type that is HER2 IHC 2+/ISH+ (excluding breast, gastric cancer, and colorectal cancer)
  Interventions: Drug: Trastuzumab deruxtecan
- Part 2 Cohort C (Experimental): HER2 IHC 2+ or 1+ endometrial cancer
  Interventions: Drug: Trastuzumab deruxtecan
- Part 2 Cohort D (Experimental): HER2 IHC 2+ or 1+ ovarian cancer
  Interventions: Drug: Trastuzumab deruxtecan
- Part 2 Cohort E (Experimental): HER2 IHC 2+ or 1+ cervical cancer
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — Trastuzumab deruxtecan by intravenous infusion
  Other Names: DS-8201a; T-DXd

SUMMARY:
This is an open-label, multi-center, multi-cohort, Phase 2 study to evaluate the efficacy and safety of trastuzumab deruxtecan (T-DXd) for the treatment of selected HER2-expressing tumors.

This study will consist of Part 1 which includes 7 cohorts of: urothelial bladder cancer, biliary tract cancer, cervical cancer, endometrial cancer, ovarian cancer, pancreatic cancer, and rare tumors; and Part 2 which includes 5 cohorts A to E of: A) any tumor type that is HER2 IHC 3+ (excluding breast, gastric cancer, and colorectal cancer), B) any tumor type that is HER2 IHC 2+/ISH+ (excluding breast, gastric cancer, and colorectal cancer), C) HER2 IHC 2+ or 1+ endometrial cancer, D) HER2 IHC 2+ or 1+ ovarian cancer, and E) HER2 IHC 2+ or 1+ cervical cancer.

Study hypothesis: Trastuzumab deruxtecan will show meaningful clinical activity and a favorable risk benefit profile in selected HER2-expressing solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced, unresectable, or metastatic disease based on most recent imaging.
* Part 1:The respective cohorts for patient inclusion are:

  * Cohort 1: Biliary tract cancer
  * Cohort 2: Bladder cancer
  * Cohort 3: Cervical cancer
  * Cohort 4: Endometrial cancer
  * Cohort 5: Epithelial ovarian cancer
  * Cohort 6: Pancreatic cancer
  * Cohort 7: Rare tumors: This cohort will consist of patients with tumors that express HER2, excluding the tumors mentioned above, and breast, non-small cell lung cancer, gastric cancer, and colorectal cancer.
* Part 2:The respective cohorts for patient inclusion are:

  * Cohort A: Metastatic or advanced solid tumors that are HER2 IHC 3+ (excluding breast, gastric cancer, and colorectal cancer). Patients with non-small cell lung cancer can be included.
  * Cohort B: Metastatic or advanced solid tumors that are HER2 IHC 2+/ISH+ any tumor type (excluding breast, gastric cancer, and colorectal cancer). Patients with non-small cell lung cancer can be included.
  * Cohort C: Metastatic or advanced solid endometrial cancer that is HER2 IHC 2+ or 1+.
  * Cohort D: Metastatic or advanced ovarian cancer that is HER2 IHC 2+ or 1+.
  * Cohort E: Metastatic or advanced solid cervical cancer that is HER2 IHC 2+ or 1+.
* Progressed following prior treatment or who have no satisfactory alternative treatment option.
* Prior HER2 targeting therapy is permitted.
* HER2 expression scored using current ASCO/CAP guidelines for scoring HER2 for gastric cancer.

  * Part 1: IHC 3+ or IHC 2+ by local or central assessment
  * Part 2: IHC and ISH results by central assessment as pre-defined for each cohort
* Has measurable target disease assessed by the Investigator based on RECIST version 1.1.
* Has protocol- defined adequate organ function including cardiac, renal and hepatic function.

Exclusion Criteria:

* History of non-infectious pneumonitis/ILD that required steroids, current ILD, or where suspected ILD that cannot be ruled out by imaging at screening
* Lung-specific intercurrent clinically significant severe illnesses
* Uncontrolled infection requiring intravenous (IV) antibiotics, antivirals, or antifungals
* Pleural effusion, ascites or pericardial effusion that requires drainage, peritoneal shunt, or Cell-free and Concentrated Ascites Reinfusion Therapy (CART
* Known Somatic DNA mutation of HER2 (ERBB2) without tumoral HER2 protein expression.
* Primary diagnosis of adenocarcinoma of the breast, adenocarcinoma of the colon or rectum, adenocarcinoma of the gastric body or gastro-esophageal junction, or non-small cell lung cancer for Part 1. For Part 2, patients with primary diagnosis of adenocarcinoma of the breast, adenocarcinoma of the colon or rectum, adenocarcinoma of the gastric body or gastro-esophageal junction will be excluded.
* Medical conditions that may interfere with the subject's participation in the study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2020-08-18 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | An average of approximately 6 months
  Confirmed ORR per RECIST 1.1 is the percentage of patients with Complete Response or Partial Response that is subsequently confirmed.

SECONDARY OUTCOMES:
Duration of response (DoR) | An average of approximately 6 months
  DOR is defined as the time from the date of first documented response until the date of documented progression or death.
Disease control rate (DCR) | An average of approximately 6 months
  DCR is the percentage of subjects who have a best overall response of complete response (CR) or partial response (PR) or stable disease (SD).
Progression free survival (PFS) | An average of approximately 6 months
  PFS is the time from date of first dose of study treatment until the date of objective disease progression or death.
Proportion of patients alive and progression-free at 6 months and 12 months | Up to 12 months
  The proportion of patients alive and progression-free at 6 and 12 months (Kaplan-Meier estimates).
Overall survival (OS) | An average of approximately 14 months
  OS is the time from date of first dose of study treatment until death due to any cause.
Proportion of patients alive at 6 and 12 months | Up to 12 months
  The proportion of patients alive at 6 and 12 months (Kaplan-Meier estimates).
Occurrence of adverse events (AEs) and serious adverse events (SAEs) | An average of approximately 8 months
  Occurrence of AEs and SAEs graded according to NCI CTCAE v5.0.
Pharmacokinetics (PK) assessed by serum concentration of T-DXd, total anti-HER2 antibody and MAAA-1181 | An average of approximately 8 months
  Individual patient data and descriptive statistics will be provided for serum concentration data at each time point for T-DXd, total anti-HER2 antibody and MAAA-1181a
The immunogenicity of T-DXd assessed by the presence of ADAs for T-DXd | An average of approximately 6 months
  Individual participant data and descriptive statistics will be provided for data at each time point.

CONTACTS AND LOCATIONS:
Locations (95):
- United States (21):
  - Research Site, Burbank, California
  - Research Site, Duarte, California
  - Research Site, Fullerton, California
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Santa Rosa, California
  - Research Site, Chicago, Illinois
  - Research Site, Muncie, Indiana
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Middletown, New Jersey
  - Research Site, Harrison, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Durham, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Seattle, Washington
- Australia (6):
  - Research Site, Auchenflower
  - Research Site, Blacktown
  - Research Site, Camperdown
  - Research Site, Heidelberg
  - Research Site, Melbourne
  - Research Site, Nedlands
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Liège
- Brazil (7):
  - Research Site, Barretos
  - Research Site, Curitiba
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, São Paulo
  - Research Site, Vitória
- Canada (7):
  - Research Site, Kelowna, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Montreal
- Czechia (5):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Prague
- India (6):
  - Research Site, Delhi
  - Research Site, Gūrgaon
  - Research Site, Kolkata
  - Research Site, Madurai
  - Research Site, Mumbai
  - Research Site, Nashik
- Italy (4):
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Roma
  - Research Site, Rome
- Japan (3):
  - Research Site, Chūōku
  - Research Site, Kashiwa
  - Research Site, Suita-shi
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Delft
  - Research Site, Groningen
- Poland (6):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Gliwice
  - Research Site, Krakow
  - Research Site, Poznan
  - Research Site, Warsaw
- Russia (3):
  - Research Site, Kaluga
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Research Site, Seoul, South Korea
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Madrid
  - Research Site, Valencia
- Taiwan (4):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (7):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Muang
  - Research Site, Ongkharak
  - Research Site, Si Sa Ket
- United Kingdom (5):
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Northwood Middlesex
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool .
  Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access.
  For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Meric-Bernstam F, Makker V, Oaknin A, Oh DY, Banerjee S, Gonzalez-Martin A, Jung KH, Lugowska I, Manso L, Manzano A, Melichar B, Siena S, Stroyakovskiy D, Fielding A, Ma Y, Puvvada S, Shire N, Lee JY. Efficacy and Safety of Trastuzumab Deruxtecan in Patients With HER2-Expressing Solid Tumors: Primary Results From the DESTINY-PanTumor02 Phase II Trial. J Clin Oncol. 2024 Jan 1;42(1):47-58. doi: 10.1200/JCO.23.02005. Epub 2023 Oct 23. PMID 37870536